CLINICAL TRIAL: NCT04014933
Title: Prospective, Non-randomised, Non-controlled Study of Reproducibility of Blood Flowmetry in Human Retina Using the Nidek Laser Speckle Flowgraphy LSFG-NAVI System
Brief Title: Reproducibility of Blood Flowmetry in Human Retina Using the Nidek Laser Speckle Flowgraphy LSFG-NAVI System
Acronym: LSFG Repro
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: LSFG Repro
Record Dates: First submitted 2019-07-03; First posted 2019-07-10 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Open Angle Glaucoma; Normal Tension Glaucoma; Healthy
Keywords: glaucoma; retinal blood flow; ocular perfusion pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- open-angle glaucoma: patients with a diagnosis of open-angle glaucoma, i.e. untreated IOP >21mmHg plus glaucomatous disc changes and/or visual field defects typical for glaucoma
  Interventions: Diagnostic Test: LASER SPECKLE FLOWGRAPHY
- normal tension glaucoma: patients with a diagnosis of normal tension glaucoma, i.e. untreated IOP </=21mmHg plus glaucomatous disc changes and/or visual field defects typical for glaucoma
  Interventions: Diagnostic Test: LASER SPECKLE FLOWGRAPHY
- healthy controls: individuals with normal optic disc and IOP </21mmHg and normal visual fields
  Interventions: Diagnostic Test: LASER SPECKLE FLOWGRAPHY

INTERVENTIONS:
Diagnostic Test: LASER SPECKLE FLOWGRAPHY — Non-invasive, real-time imaging and measurement of ocular blood flow of the optic disc and peripapillary region

SUMMARY:
In addition to intraocular pressure blood perfusion pressure in the optic nerve is an important factor determing the cause of glaucoma. Increasing evidence suggests that in glaucoma patients retinal blood may be decreased.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO) glaucoma is the second leading cause of blindness. Glaucoma is a global problem, which is becoming even more important as the human life expectancy increases. Although the causes of glaucoma are uncertain, mainly intraocular pression (IOP), genetics, and ocular blood perfusion pressure in the optic nerve determine the cause of the disease. Increasing evidence suggests that in glaucoma patients retinal blood flow is decreased leading to progression and to damage of the optic nerve.

In order to measure the peripapillary blood flow a variety of devices using different techniques of flowmetry have been developed. In this study, the reproducibility of the retinal flowmetry measured with the LSFG-NAVI device from Nidek will be investigated. A high reproducibility is crucial for the clinical value of any measuring device.

ELIGIBILITY:
Inclusion Criteria:

* signed Patient Informed Consent form
* Be at least 18 years old
* Diagnosis of primary or secondary open-angle glaucoma or normal tension glaucoma or healthy controls

Exclusion Criteria:

* Age < 18 years
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* No vulnerable participants will be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3 groups as described above will be recruted from the outpatient department of the Ophthalmology Department at the UniversityHospital Zurich, Zurich, Switzerland and the Ophthalmology Department at the Cantonal Hospital Aarau, Aarau, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Coefficients of variation (COV) | 1 month
  COVs from 3 measurements of ocular blood flow at visit 1 of observer 1 and at visit 1 of observer 1 and from observer 2 will be computed.
intraclass correlation coefficients (ICCs) | 1 month
  Intraobserver ICC, interobserver ICC, and inter-session ICC will be computed

SECONDARY OUTCOMES:
Cofounder | 1 month
  Blood pressure will be checked as potential cofounder
Cofounder | 1 month
  heart rate will be checked as potential cofounder
Cofounder | 1 month
  spherical equivalent will be checked as potential cofounder
Cofounder | 1 month
  intraocular pressure will be checked as potential cofounder

CONTACTS AND LOCATIONS:
Overall Officials: Marc Töteberg-Harms, MD, FEBO, Principal Investigator — UniversityHospital Zurich, Department of Ophthalmology, Zurich, Switzerland
Locations (1):
- Department of Ophthalmology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No